CLINICAL TRIAL: NCT05511103
Title: A Cohort of Acute, Ischemic and Rare Neuropathies
Acronym: CAIRN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CAIRN
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Neuropathy; Rare Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuropathies are defined as the clinical, electrical, biological and histological manifestations of peripheral neuron damage. They represent a heterogeneous group of disorders and are responsible for disabling sensory and motor disorders. Their diagnosis is based on a set of clinical arguments confirmed by the electromyogram. This allows to specify the site of the damage, its severity, and to follow the evolution of the disease.

To date, the diagnosis of peripheral nerve injury secondary to occlusion of arterial trunks is rarely evoked; its clinical, electromyographic and prognostic characteristics are poorly known. Indeed, the rare cases reported in the literature are from vascular specialties, with little data on neurological symptoms, neurophysiological diagnostic elements and prognosis.

However, these unrecognized and underdiagnosed neuropathies are sometimes indicative of severe vascular damage for which urgent management is necessary. Neurological symptoms should then be treated as warning signs and the correct recognition of the early ischemic vascular etiology may lead to an optimized medical management.

The objectives of this study will be to describe the clinical presentation of these neuropathies, to discuss their electrophysiological diagnostic characteristics, to compare the demographic data with those from the literature, and to evaluate the functional prognosis of these attacks. A better knowledge of this rare etiology of neuropathy would allow to better inform the patients and to optimize the diagnostic and therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient hospitalized or seen in neurophysiological consultation/exploration in the Neurology Department within the Groupe Hospitalier Paris Saint-Joseph
* Diagnosis of acute or subacute peripheral nerve ischemia
* French speaking patient

Exclusion Criteria:

* Patient with impaired comprehension making it impossible to understand the protocol
* Patient under guardianship or curatorship
* Patient under court protection
* Patient deprived of liberty
* Patient or relative who objects to the use of his/her data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized or seen in neurophysiological consultation/exploration in the Neurology Department within the Groupe Hospitalier Paris Saint-Joseph, with Diagnosis of acute or subacute peripheral nerve ischemia
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of patients according to their neurophysiological impairment | Month 1
  This outcome corresponds to the description of patient demographics and cardiovascular history/risk factors.

SECONDARY OUTCOMES:
Prognostic factors for functional recovery | Month 1
  This outcome corresponds to the the prognosis of the disease (return to the previous state/persistence of a partial deficit/persistence of symptoms) and the time to improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Roubeau, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Siao P, Kaku M. A Clinician's Approach to Peripheral Neuropathy. Semin Neurol. 2019 Oct;39(5):519-530. doi: 10.1055/s-0039-1694747. Epub 2019 Oct 22. PMID 31639835
- [Background] Abdellaoui A, West NJ, Tomlinson MA, Thomas MH, Browning N. Lower limb paralysis from ischaemic neuropathy of the lumbosacral plexus following aorto-iliac procedures. Interact Cardiovasc Thorac Surg. 2007 Aug;6(4):501-2. doi: 10.1510/icvts.2007.151993. Epub 2007 Apr 17. PMID 17669917
- [Background] Abdelhamid MF, Sandler B, Awad RW. Ischaemic lumbosacral plexopathy following aorto-iliac bypass graft: case report and review of literature. Ann R Coll Surg Engl. 2007 Jul;89(5):W12-3. doi: 10.1308/147870807X188470. PMID 17688710
- [Background] Deylgat B, Wallaert P, De Smul G, Van Lysebeth L, Ceuppens H. Unilateral lower limb paralysis after aortobifemoral bypass graft for ruptured abdominal aortic aneurysm: a case report. Vasc Endovascular Surg. 2009 Dec;43(6):606-9. doi: 10.1177/1538574409345032. Epub 2009 Oct 14. PMID 19828587
- [Background] Winston P, Bakker D. Ischemic Monomelic Neuropathy: The Case for Reintroducing a Little-Known Term. Can J Neurol Sci. 2020 Sep;47(5):697-699. doi: 10.1017/cjn.2020.88. Epub 2020 May 4. PMID 32362289